CLINICAL TRIAL: NCT05159037
Title: Using the Musical Track From Gaze-Contingent Music Reward Therapy as a Treatment Booster in Stressful Situations Among Highly Socially Anxious Participants
Brief Title: Using the Musical Track From GC-MRT as a Treatment Booster in Stressful Situations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAUgcMRTbooster
Record Dates: First submitted 2021-11-15; First posted 2021-12-15 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Social Anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active GC-MRT Booster (Experimental): Following four sessions of Gaze-Contingent Music Reward Therapy training participants' attention away from threats and towards neutral stimuli, participants will listen to a musical track they will have been trained with prior to a stressful speech task.
  Interventions: Behavioral: Gaze Contingent Music Reward Therapy; Behavioral: Music Booster
- Control Booster (Placebo Comparator): Following four sessions of Gaze-Contingent Music Reward Therapy training participants' attention away from threats and towards neutral stimuli, participants will listen to a musical track they will not have been trained with but ranked as highly liked prior to a stressful speech task.
  Interventions: Behavioral: Gaze Contingent Music Reward Therapy; Behavioral: Music Booster

INTERVENTIONS:
Behavioral: Gaze Contingent Music Reward Therapy — Feedback according to participants' viewing patterns, in order to modify their attention.
Behavioral: Music Booster — Participants listen to a musical track they ranked as highly liked before a stressful situation

SUMMARY:
The study examines whether musical tracks played during gaze contingent music reward therapy (GC-MRT) for social anxiety could later be used as a booster to reduce anxiety before a stressful situation. To this end, highly socially anxious participants will undergo 4 GC-MRT sessions designed to train participants' attention away from threat and towards neutral social stimuli. Subsequently, participants will be asked to perform a socially stressful speech task. Prior to the speech, half of the participants will listen to a musical track the participants were trained with, and half of the participants will listen to a musical track the participants like but were not trained with during the GC-MRT sessions. The investigators expect that listening to musical track taken from the GC-MRT sessions will moderate the increase in anxiety levels prior to the speech and will improve performance during the speech compared to a non-trained musical track.

DETAILED DESCRIPTION:
Gaze contingent music reward therapy (GC-MRT) is designed to modify threat-related attention biases through operational conditioning between beloved music and gaze patterns favoring neutral stimuli over threat-related stimuli. GC-MRT has shown efficacy in reducing social anxiety symptoms. The current study is designed to explore whether the musical tracks played during the GC-MRT conditioning could be later used as a treatment booster to reduce anxiety in a socially stressful situation. To this end, 60 high socially anxious participants will undergo four GC-MRT sessions and then will be asked to perform a stressful speech task. Prior to the speech, half of the participants (randomly determined) will listen to a musical track the participants were trained with, and half of the participants will listen to a musical track the participants like but were not trained with during GC-MRT sessions. The investigators expect that the listening to musical track taken from the GC-MRT sessions will moderate the increase in anxiety levels prior to the speech and will improve performance during the speech compared to a non-trained musical track.

ELIGIBILITY:
Inclusion Criteria:

* a signed consent form
* an age of 18 years or above
* a score greater than 60 on LSAS

Exclusion Criteria:

* a self-reported history of neurological or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-07 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline - the Liebowitz Social Anxiety Scale - Self Reported Version | 2 days before intervention, 4-10 days after intervention completion
  The LSAS is a 24-item scale, each item corresponding to a situation selected on the basis of clinical experience. Each item is rated on a severity scale ranging from 0 to 3 with regard to the passing week, measuring separately two components of social anxiety, specifically, fear/anxiety and avoidance of social interaction and performance situations.
Change from baseline - the Visual Analogue Scale - Anxiety | 4-10 days after intervention completion (baseline of the speech session, after introducing the speech task, after listening to a musical track, after preparation to the speech,after the speech is over).
  The Visual Analogue Scale Anxiety (VAS-A) measures state anxiety. Participants are instructed to use the computer mouse and place the locator at the scale position representing their current level of anxiety in response to the question, "How anxious do you feel right now?". The VAS is divided into thirty units from 0 ("calm") to 30 ("anxious") while the participants do not see the division into calves and are asked to answer according to their feeling.

SECONDARY OUTCOMES:
PSPS (Public Speaking Performance Scale) | 4-10 days after intervention completion (During speech task)
  The Public Speaking Performance Scale comprises 17 items concerning speech quality. Items are rated by independent judges on a 5-point scale from 0 (not at all) to 4 (very much). Higher scores denote worse performance.

OTHER OUTCOMES:
Change from baseline - viewing patterns on threat-neutral face matrices | At the first day of intervention, 4-10 days after intervention completion
  Gaze patterns, and specifically attention allocation to threat will be used as moderators for clinical outcome, as well as indicators of target engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT05159037/SAP_000.pdf